CLINICAL TRIAL: NCT07274085
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic (PK) Characteristics, and Preliminary Antitumor Efficacy of HDM2017 in Participants With Advanced Malignant Solid Tumors
Brief Title: A Phase 1 Study of HDM2017 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDM2017-101
Record Dates: First submitted 2025-11-24; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HDM2017 (Experimental): Participants will receive escalating doses of HDM2017, then at least 2 dose levels will be selected for dose expansion to determine the RP2D
  Interventions: Drug: HDM2017

INTERVENTIONS:
Drug: HDM2017 — Participants will be treated with HDM2017 intravenous infusion

SUMMARY:
This is a phase I clinical study. All subjects are patients with advanced solid tumors. The purpose of this study is to to evaluate the safety, tolerability, pharmacokinetic (PK) characteristics, and preliminary antitumor efficacy of HDM2017 in patients with advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide written informed consent.
2. Male or female participants aged 18 to 75 years.
3. Participants with histologically or cytologically confirmed locally advanced unresectable or metastatic malignant solid tumors who have failed adequate standard of care, or are intolerant to standard of care, or have no effective standard treatment options.
4. Be able to provide archived tumor tissue during the screening period.
5. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
6. Life expectancy ≥3 months.
7. According to RECIST v1.1, participants must have at least one measurable lesion.
8. Has adequate organ function.
9. All subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 7 months after the last dose of study treatment.
10. Be willing and able to complete regular visits, treatment plans, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Participants who have previously received ADC therapy containing Top I inhibitors, or other drug therapy targeting the CDH17 target.
2. Participants who have received the following treatments:

   1. Participants who have undergone major surgery within 4 weeks before the first dose;
   2. Participants who have received radiotherapy involving the bone marrow or extensive radiotherapy within 4 weeks before the first dose; or local radiotherapy within 2 weeks before the first dose;
   3. Participants receiving continuous systemic corticosteroid therapy;
   4. Participants who have received systemic antitumor therapy, or any other investigational drug therapy within 4 weeks or 5 half-lives (whichever is shorter; at least 2 weeks) before the first dose.
3. Participants with other malignant tumors within the past 5 years, other than the tumor being treated in this study, with the exception of locally cured tumors (such as basal cell carcinoma, cutaneous squamous cell carcinoma, superficial bladder cancer, carcinoma in situ of the cervix or breast).
4. Related AEs from prior therapy (except for alopecia and ≤Grade 2 sensory neuropathy) have not recovered to ≤Grade 1 or baseline level.
5. Known weight loss of >10% within 2 months before the first dose of study drug or other indicators showing severe malnutrition.
6. History of gastrointestinal perforation, abdominal fistula, or extensive intestinal resection within 6 months before the first dose; complete or incomplete gastrointestinal obstruction or intra-abdominal abscess within 3 months before the first dose.
7. History of gastrointestinal hemorrhage within 3 months before the first dose, or a clear gastrointestinal hemorrhagic diathesis.
8. Participants with known active CNS metastasis.
9. Participants with cardiovascular/cerebrovascular disorder, symptoms, or manifestations.
10. Participants with active syphilis, history of human immunodeficiency virus (HIV) infection, active hepatitis B virus (HBV) or active hepatitis C virus (HCV), except for asymptomatic chronic hepatitis B or C virus carriers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 30 days after the last dose of IMP
  The MTD will be determined using DLTs
Recommended Phase 2 Dose (RP2D) | 30 days after the last dose of IMP
  The RP2D will be determined using dose limiting toxicities (DLTs) and all other available study data
Type, incidence and severity of Adverse Events | 30 days after the last dose of IMP
  Safety and tolerability profile assessed by the Common Terminology Criteria for Adverse Events v5.0

SECONDARY OUTCOMES:
Tmax | 30 days after the last dose of IMP
  Time to reach the maximum blood concentration
Cmax | 30 days after the last dose of IMP
  Maximum observed blood concentration
Incidence of anti-drug antibody (ADA) | 30 days after the last dose of IMP
  The proportion of patients with positive ADA results
Objective Response Rate (ORR) | 30 days after the last dose of IMP
  ORR is defined as the proportion of subjects with BOR response of CR or PR (based on RECIST Version 1.1).
Disease control rate (DCR) | 30 days after the last dose of IMP
  DCR is defined as the proportion of subjects with response of CR, PR and SD (based on RECIST Version 1.1).
Duration of Response (DoR) | 30 days after the last dose of IMP
  The time from first documented evidence of CR or PR until time of first documented disease progression.
Progression Free Survival (PFS) | 30 days after the last dose of IMP
  PFS is defined as the interval between first dose and the earliest date of disease progression or death due to any cause.
Overall survival (OS) | 30 days after the last dose of IMP
  OS is defined as the time from first dose until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No